CLINICAL TRIAL: NCT01488214
Title: Assessment of Neuropsychiatric Involvement in Systemic Sclerosis.
Brief Title: Neuropsychiatric Scleroderma Study: Systematic Evaluation of Neuropsychiatric Involvement in Systemic Sclerosis
Acronym: NeuroScS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009_10; PHRC 2009/API (Other: DHOS); 2009-A01313-54 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2011-11-25; First posted 2011-12-08 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis; neuropsychiatric manifestations; magnetic resonance imaging
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Magnetic Resonance Spectroscopy; Psychiatry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scleroderma patient (Experimental): Evaluation of Scleroderma patient
  Interventions: Other: Magnetic resonance Imaging
- Healthy subjects (Placebo Comparator): Evaluation of healthy subjects
  Interventions: Other: Magnetic resonance Imaging

INTERVENTIONS:
Other: Magnetic resonance Imaging — Magnetic resonance Imaging Assessment
  Other Names: Cognitive, psychiatric and neurological evaluation

SUMMARY:
Systemic sclerosis is a rare disease with vascular involvement and systemic fibrosis. This disease is usually thought to spare central nervous system. However, neuropsychiatric manifestations like depression and cognitive functions impairment seem to be frequent. Pathophysiology of this neuropsychiatric manifestations is currently unknown. White matter hyperintensities have been reported suggested CNS vascular manifestations in systemic sclerosis. Whether this CNS vascular involvement plays a role in neuropsychiatric manifestations in systemic sclerosis is unknown. The primary objective of this prospective and multicentre study is to assess a link between neuropsychiatric manifestations and CNS involvement in systemic sclerosis. Secondary objectives are to assess the frequency of neuropsychiatric manifestations, to compare central nervous system abnormality between scleroderma patient and healthy subjects. Central nervous system involvement and neuropsychiatric manifestations will be systematically assessed through central nervous system imaging and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 yo
* With scleroderma (American College of Rheumatology and/or Leroy et Medsger)
* Informed consent given

Exclusion Criteria:

* Other auto-immune disease
* non french native speakers
* severe arterial hypertension
* diabetes
* anemia
* renal insufficiency
* cranial trauma
* history of neurological disorder or neurotoxic treatment
* pregnancy or breast feeding
* impossibility or non compliance to perform the protocol flow chart
* contra indications to MRI

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Odds-ratio between neuropsychiatric manifestations and magnetic resonance imaging abnormalities | 5 weeks
  Odds-ratio between neuropsychiatric manifestations and magnetic resonance imaging abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD, PhD, Study Chair — Lille University Hospital; Amar Smail, MD, Principal Investigator — Amiens University Hospital; Boris Bienvenu, MD, PhD, Principal Investigator — University Hospital, Caen; Isabelle Marie, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - Caen University Hospital, Caen, Calvados
  - Lille University hosiptal, Lille, Nord
  - Rouen University hospital, Rouen, Seine-Maritime
  - Amiens Launay, Amiens, Sommes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Launay D, Remy-Jardin M, Michon-Pasturel U, Mastora I, Hachulla E, Lambert M, Delannoy V, Queyrel V, Duhamel A, Matran R, De Groote P, Hatron PY. High resolution computed tomography in fibrosing alveolitis associated with systemic sclerosis. J Rheumatol. 2006 Sep;33(9):1789-801. PMID 16960939
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/16960939